CLINICAL TRIAL: NCT02630602
Title: Functional Goat Cheese Effect in Lipid Profile Change
Acronym: LODYN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LODYN 4092
Record Dates: First submitted 2015-12-11; First posted 2015-12-15 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Obesity and Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Functional goat cheese (Active Comparator): The functional cheese is rich in conjugated linoleic acid (CLA) and omega-3. It was used for obese and overweight people, who need a special diet advice to control of lipid profile. 9,3% of polyunsaturated fatty acids 60 g per day during 12 weeks
  Interventions: Dietary Supplement: Functional goat cheese
- Control cheese (Placebo Comparator): Control cheese, not enriched with conjugated linoleic acid (CLA) and omega-3 4.1% of polyunsaturated fatty acids. 60 g per day during 12 weeks
  Interventions: Dietary Supplement: Control cheese

INTERVENTIONS:
Dietary Supplement: Functional goat cheese — 60 g per day during 12 weeks
  Arms: Functional goat cheese
Dietary Supplement: Control cheese — 60 g per day during 12 weeks
  Arms: Control cheese

SUMMARY:
The purpose this study was to evaluate the therapeutic effect of a functional goat cheese on obese and overweight people with altered lipid profile. The functional goat cheese containing polyunsaturated fatty acid, in amounts exceeding other cheese, was developed to benefit cardiovascular health of people who need to normalize lipid profile; which in the long term can contribute to the prevention of cardiovascular diseases.

DETAILED DESCRIPTION:
A randomized, parallel, double-blind, controlled is being performing to evaluate the effect of a functional goat cheese on lipid profile in overweight or obese volunteers who need a special diet.

Were included 60 volunteers (men and women) aged between 18 and 65 years (IMC ≥27<40 Kg/m2) with a cardiovascular risk (<10%). The volunteers are being followed at La Paz University Hospital of Madrid. For 12 weeks, the volunteers should consume 60 g of cheese daily (functional cheese or control cheese) and to receive advice to follow a balanced and individualized hypocaloric diet as well as physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers with overweight type II or obesity type I or II (IMC ≥27<40 Kg/m2).
* Cardiovascular risk < 10% and almost two of follow factors:

Men ≥ 45 years old or women ≥ 55 years old; Familiar background of premature cardiovascular disease; HDL cholesterol <40 mg/dL for men and <50 mg/dL for women; Total cholesterol ≥ 200 mg/dL; Triglycerides ≥ 150 mg/dL and < 200 mg/dL; LDL ≥ 130 mg/dL and < 160 mg/dL; Smoker

* Accept advises to perform a balanced hypocaloric diet and regular practice of physical activity.
* Signed informed consent.

Exclusion Criteria:

* Individuals with Diabetes Mellitus type 1;
* Individuals with Diabetes Mellitus type 2, using medication;
* Individuals with Dyslipidemia, using drug;
* Individuals with high blood pressure, using medication;
* Individuals with allergies to dairy protein;
* Individuals with severe diseases (hepatic, kidney, cancer…);
* Individuals with drugs or supplements consumption to weight lost;
* Individuals that consume drugs, ω-3 supplements or supplement that can modify the lipid and / or glucose profile (statins, fibrates, diuretics, corticosteroids, insulin…);
* Individuals who have participated in programs and / or clinical trials of weight control in the last 6 months;
* Individuals with increased alcohol consumption 30g/day;
* Individuals that stop smoking in the next 20 weeks (during the study);
* Individuals with mental disease or low cognitive function;
* Pregnant women or breastfeeding;
* Individuals with intensive physical activity;
* Individuals with physical problems complying with the recommendations of physical activity and diet general recommendations.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
change from baseline total cholesterol | 0 and 12 weeks
change from baseline Low density lipoprotein cholesterol | 0 and 12 weeks
change from baseline High density lipoprotein cholesterol | 0 and 12 weeks

SECONDARY OUTCOMES:
change from baseline Triglycerides | 0 and 12 weeks
change from baseline Apolipoprotein A1 | 0 and 12 weeks
change from baseline Apolipoprotein B | 0 and 12 weeks
change from baseline Free fatty acids (FFA) in the plasma | 0 and 12 weeks
change from baseline Erythrocyte membrane fatty acid composition | 0 and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Gomez, MD. PhD, Principal Investigator — HOSPITAL LA PAZ
Locations (1):
- La Paz University Hospital, Madrid, Madrid, Spain